CLINICAL TRIAL: NCT01615302
Title: Use of Platelet Rich Plasma (PRP) as an Adjunct in the Treatment of High Peri-anal Fistulas.
Brief Title: Is the Use of Blood Platelets Effective in the Treatment of Difficult Fistulas Related to the Anal Sphincter?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Biomet Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC 10-1-082
Record Dates: First submitted 2012-05-30; First posted 2012-06-08 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Rectal Fistula
Keywords: Rectal Fistula; Peri-anal Fistula; Platelet-Rich Plasma; Mucosa advancement flap
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mucosa advancement flap (Active Comparator)
  Interventions: Procedure: Mucosa advancement flap
- Mucosa advancement flap + PRP (Experimental): Platelet rich plasma added to the mucosa advancement flap
  Interventions: Procedure: Mucosa advancement flap; Other: Platelet rich plasma (PRP)

INTERVENTIONS:
Procedure: Mucosa advancement flap — Mucosa advancement flap will be performed at the starting point of the fistula in the rectum
Other: Platelet rich plasma (PRP) — The PRP will be injected into the fistula, after the mucosa advancement flap was created.
  For the PRP we will need to take 55 millilitres of blood of the patient. This blood will be centrifuged into PRP.
  Arms: Mucosa advancement flap + PRP

SUMMARY:
Rationale:

Closure of the internal opening is the most accepted standard procedure in the treatment of peri-anal fistulas. The mucosal advancement flap is considered as golden standard. In one out of the three patients mucosal flap repair fails. Possible causal factors are incomplete clearance of pus and debris, incomplete closure of the internal opening, inappropriate host response in patients with risk factors like smoking or diabetes. Platelet derived growth factors may facilitate closure of the internal opening, especially in patients with impaired wound healing.

Objective:

The use of autologous platelet rich plasma (PRP) as an adjunct to the staged mucosal advancement flap to achieve a better closure rate of complex peri-anal fistula's.

Study design:

Randomized, multicenter trial.

Study population:

Patients with complex cryptoglandular peri-anal fistula's.

Intervention:

Injection of PRP in the curretted fistula track under the mucosal flap.

Main study parameters/endpoints:

* Recurrence rate
* Post-operative pain
* Continence
* Quality of life.

Nature and extent of the burden and risks associated with participation, group relatedness:

Because autologous blood is used, no extra risk are expected.

ELIGIBILITY:
Inclusion Criteria:

* Complex peri-anal fistula.
* Able to understand informed consent.

Exclusion Criteria:

* Pregnancy
* Local malignancy
* Crohn's disease or Ulcerative colitis
* Traumatic or iatrogenic lesion
* Thrombocytopenia
* Splenomegaly
* Bleeding disorders
* Hematologic malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of fistulas | Assessed up to 104 weeks after operation
  The surgeon or docter in the outpatient clinic will decide if there is a recurrent fistula or not.
  In case of doubt a MRI will be made.

SECONDARY OUTCOMES:
Pain | Assessed at 2 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Quality of Life | Assessed at 2 weeks after operation
  Measured using the SF-36v2 questionnaire
Incontinence | Assessed at 2 weeks after operation
  Measured using the Vaizey score
Pain | Assessed at 4 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Pain | Assessed at 16 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Pain | Assessed at 24 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Pain | Assessed at 52 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Pain | Assessed at 104 weeks after operation
  Measured using the Visual Analogue Scale (VAS-score)
Quality of life | Assessed at 4 weeks after operation
  Measured using the SF-36v2 questionnaire
Quality of Life | Assessed at 16 weeks after operation
  Measured using the SF-36v2 questionnaire
Quality of life | Assessed at 24 weeks after operation
  Measured using the SF-36v2 questionnaire
Quality of life | Assessed at 52 weeks after operation
  Measured using the SF-36v2 questionnaire
Quality of life | Assessed at 104 weeks after operation
  Measured using the SF-36v2 questionnaire
Incontinence | Assesed at 4 weeks after operation
  Measured using the Vaizey score
Incontinence | Assessed at 16 weeks after operation
  Measured using the Vaizey score
Incontinence | Assessed at 52 weeks after operation
  Measured using the Vaizey score
Incontinence | Assessed at 24 weeks after operation
  Measured using the Vaizey score
Incontinence | Assessed at 104 weeks after operation
  Measured using the Vaizey score

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie O. Breukink, MD, PhD, Principal Investigator — Maastricht University Medical Center; Cor G.M.I. Baeten, MD, PhD, Prof., Study Director — Maastricht University Medical Center
Locations (6):
- Netherlands (6):
  - Atrium Medisch Centrum, Heerlen, Limburg
  - University Hospital Maastricht, Maastricht, Limburg
  - Laurentius ziekenhuis, Roermond, Limburg
  - Amphia ziekenhuis, Breda, North Brabant
  - Catharina ziekenhuis, Eindhoven, North Brabant
  - Refaja Ziekenhuis, Stadskanaal, Provincie Groningen

REFERENCES:
- [Background] van der Hagen SJ, Baeten CG, Soeters PB, van Gemert WG. Autologous platelet-derived growth factors (platelet-rich plasma) as an adjunct to mucosal advancement flap in high cryptoglandular perianal fistulae: a pilot study. Colorectal Dis. 2011 Feb;13(2):215-8. doi: 10.1111/j.1463-1318.2009.01991.x. PMID 19575739
- [Derived] Gottgens KW, Vening W, van der Hagen SJ, van Gemert WG, Smeets RR, Stassen LP, Baeten CG, Breukink SO. Long-term results of mucosal advancement flap combined with platelet-rich plasma for high cryptoglandular perianal fistulas. Dis Colon Rectum. 2014 Feb;57(2):223-7. doi: 10.1097/DCR.0000000000000023. PMID 24401885